CLINICAL TRIAL: NCT02861144
Title: Partnerships for Cardiometabolic Disparities in Native and Pacific People
Brief Title: The Hanapū Study: Incentivized Partnerships to Reduce Diabetes Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHS#18539; 3P20MD000173-09S1 (NIH)
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Other): Patient participants in the intervention arm will receive diabetes self-management program, Ma ka hana ka ̒ike which includes 5 interactive group sessions lasting 1-1/2 hours in length delivered by community peer educators once a month for 4.5 months. After 4.5 months, the patient will receive 4 monthly boosters by mail that will reinforce information from the Ma ka hana ka ̒ike program. Completion of diabetes process and glycemic outcomes will trigger the modest financial incentives.
  Health care provider participants in the intervention arm will receive educational resources, Hanapū Provider Toolbox to guide their patients to optimal glycemic control.They will receive modest financial incentives when their patients complete clinical tests and achieve glycemic target.
  Interventions: Other: Ma ka hana ka ̒ike; Other: Hanapū Provider Toolbox
- Usual Care (No Intervention): Patient participants in the usual care arm will receive 5 mail-out diabetes self management education booklets endorsed by the American Diabetes Association (ADA) and the National Institute for Diabetes, Digestive and Kidney disease for 4.5 months. Patients will see their doctor according to usual care practice. After 4.5 months, the patients will receive 4 monthly boosters in mail reinforcing the previous mail-out diabetes self-management program materials.
  Health care provider participants in the usual care arm will receive the latest ADA guidelines to use in their treatment plan of their patients.

INTERVENTIONS:
Other: Ma ka hana ka ̒ike — Ma ka hana ka ̒ike is a self-management program for diabetic patients which includes 5 interactive group sessions lasting 1-1/2 hours in length delivered by community peer educators once a month for 6 months.
  Arms: Intervention
Other: Hanapū Provider Toolbox — Hanapū Provider Toolbox is an educational tools that will aid the health care providers in guiding their patients to optimal glycemic control.
  Arms: Intervention

SUMMARY:
The Hanapū Study: Incentivized Partnerships to Reduce Diabetes Disparities is a randomized control trial that will test the effectiveness of partnership incentives plus evidence-based education to optimize glycemic outcomes among diabetic patients compared with usual care.

DETAILED DESCRIPTION:
The Hanapū Study will use a block randomization study design to enroll 100 diabetic patients in each arm (n = 200) followed over 9 months. Providers will identify diabetic patients. After the baseline visit is completed, patient(s) and their provider will be randomized to either Intervention or Usual care arm as partners. The intervention arm will receive diabetes self-management education and modest financial incentives (gift cards) for completing diabetes process and glycemic outcomes according diabetes "best practices". Usual care patients will receive an equal number of educational materials on diabetes self-management via mail and will receive usual care through their provider but will not receive additional incentives for reaching glycemic outcomes. Both arms of the study will complete outcome visits at baseline, 4.5 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of diabetes mellitus
* HbA1c >7%
* Not planning to move out of the State
* Able to fully participate in either intervention or usual care arms.

Exclusion Criteria:

* Pregnancy
* End Stage Renal Disease requiring dialysis
* Any medical condition that would prevent participation in all aspects of the study protocol (including major psychiatric diagnosis) or with < 6 month expected survival, as determined by the patient's physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c | Baseline, 4.5 months and 9 months
  HbA1c assessment will be done at baseline and during the intervention follow up periods (4.5 and 9 months) to see incremental improvement (0.5% decrease in HbA1c) or achieving optimal control (HbA1c < 7%).

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie K Mau, MD, Principal Investigator — The University of Hawaii

IPD SHARING:
Plan to Share IPD: No